CLINICAL TRIAL: NCT04171609
Title: Expressive Writing for Resilience in Adult Cancer Survivors.
Brief Title: Expressive Writing for Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00101278
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2019-11

CONDITIONS: Cancer Survivors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer survivors (Experimental): Adult survivors of any kind of cancer (except for minor skin cancer) are eligible to participate
  Interventions: Behavioral: Expressive writing

INTERVENTIONS:
Behavioral: Expressive writing — During this daylong expressive writing workshop intervention, the writing instructor coached participants through a series of simple writing exercises. Participation required neither any prior writing experience, nor any desire to become a writer. The practices cultivate natural abilities to express the ideas that define who you are and how you experience your life.

SUMMARY:
The purpose of this study is to determine whether a 1-day expressive writing intervention for adult cancer survivors improves resilience scores as measured by the Connor-Davidson Resilience Scale (CD-RISC).

DETAILED DESCRIPTION:
The purpose of this study is to determine whether a 1-day expressive writing intervention for adult cancer survivors improves resilience scores as measured by the Connor-Davidson Resilience Scale (CD-RISC).

ELIGIBILITY:
Inclusion Criteria:

* Have ever received a cancer diagnosis
* Have completed cancer treatment (e.g., surgery, radiation, or chemotherapy)
* Are able to speak, read, write, and understand English
* Are cognitively able to provide consent
* Are able to travel to Durham to participate in the 1-day writing intervention

Exclusion Criteria:

-Cancer diagnosis was skin cancer that did not require additional treatment after surgical removal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Change in resilience as measured by the Connor-Davidson Resilience Scale | Baseline, 6 months
  This 25-item scale addresses resilience, and has been studied in a variety of populations. Resilience is considered as the capacity to overcome adversity.

SECONDARY OUTCOMES:
Post-writing survey | 1 day (collected during the 1-day intervention)
  This five-question survey is used after each writing exercise to measure how respondents reflect on their writing. This survey asks participants to respond to the first four questions using a 10-point Likert-type scale endorsing the degree to which each item reflects their thoughts and feeling about their writing. The fifth question asks for a free-response reflection on how they think and feel about how their writing went.
Change in quality of life as measured by the Quality of Life Patient/Cancer Survivor Version (QOL-CSV) | Baseline, 6 months
  The QOL-CSV is a 41-item ordinal scale measuring quality of life as a cancer patient that originated in use for pain research and was recently adapted for use in long-term cancer survivorship. This survey asks participants to measure their quality of life in terms of the physical, psychological, social, and spiritual dimensions of well-being.
Change in perceived stress as measured by Perceived Stress Scale (PSS-10) | Baseline, 6 months
  The PSS-10 is a well-known 10-item questionnaire used to evaluate responders' perceptions about their level of stress and their ability to cope with stress over the last month. Results from this questionnaire have demonstrated acceptable levels of validity and reliability. This inventory asks participants to respond using a 10-point Likert-type scale when endorsing the degree to which each item best reflects their thoughts and feelings within the past month.
Change in depression as measured by Center for Epidemiological Studies Depression Scale Revised (CESD-R) | Baseline, 6 months
  The 20-item CESD-R is one of the most common screening tests that measures depressive feelings and behaviors within the past week.
Qualitative follow-up questionnaire | 6 months
  This qualitative follow-up questionnaire will be administered 6 months after the study intervention to capture participants' reflections on their experience in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Glass, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Integrative Medicine, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No